CLINICAL TRIAL: NCT01944059
Title: The Role of Theramine® in the Prevention of Migraine Headache: A Pilot Study
Brief Title: Theramine® in the Prevention of Migraine Headache
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding Discontinued
Sponsor: Vincent Martin, MD (Industry)
Collaborators: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor-Investigator, Vincent Martin, MD, Vincent Martin MD, University of Cincinnati Physicians Company, Targeted Medical Pharma
Organization: Targeted Medical Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VM-2013-001
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Migraine Headaches
MeSH Terms: conditions — Migraine Disorders | interventions — Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theramine (Active Comparator): 2 capsules before breakfast and dinner (BID) for 16 weeks.
  Migraine preventative medications will be permitted, but no changes in dosage will be allowed during the four month study. Migraine abortive meds will be permitted and will be administered per their standard routine.
  Interventions: Drug: Theramine (medical food/old drug)
- placebo (l-alanine) (Placebo Comparator): 2 capsules before breakfast and dinner (BID) for 16 weeks.
  Migraine preventative medications will be permitted, but no changes in dosage will be allowed during the four month study. Migraine abortive meds will be permitted and will be administered per their standard routine.
  Interventions: Other: Placebo (l-alanine)

INTERVENTIONS:
Drug: Theramine (medical food/old drug) — Theramine® is a prescription medical food that is composed of variety of amino acids and/or their precursors.
  Arms: Theramine
Other: Placebo (l-alanine) — Theramine like placebo comparator
  Arms: placebo (l-alanine)

SUMMARY:
The purpose of this study is to evaluate the efficacy of Theramine® as a preventative for migraine headaches.

DETAILED DESCRIPTION:
This randomized double blind placebo-controlled study will enroll approximately 80 otherwise healthy subjects with a diagnosis of migraine headache. All subjects will be medically stable at enrollment and be on a stabilized dosage of daily medications.

The study duration will be approximately four months and the study will be divided into 3 phases (described below). Participants will complete daily headache diaries throughout all phases of the study, which will assess the presence or absence of headache as well as its characteristics (e.g. unilateral vs. bilateral, worse with exertion, moderate to severe intensity, throbbing quality, presence of associated symptoms [nausea, vomiting, photophobia, phonophobia]. The peak severity of the headaches will also be rated on a 0-10 scale each day. The characteristics of the headaches will enable us to classify headache days into those with migraine and non-migraine headaches. A migraine day will be considered any day with a moderate to severe headache that has one of the following two associated symptoms: 1) both photophobia and phonophobia or 2) nausea or vomiting. A headache day will be defined as the presence of any headache regardless of its characteristics.

Migraine preventative medications will be permitted, but no changes in dosage will be allowed during the four month study. Migraine abortive meds will be permitted and will be administered per their standard routine.

Phase 1: During this phase, participants will complete daily headache diaries for 30 days, but no study medication will be given. This phase will last approximately 1 month and will establish a baseline for the frequency of migraine in the absence of study medication.

Phase 2: Phase 2 will last for 1 month and represents the time period of initiation of the study medication. Participants will be randomized to either 2 capsules of Theramine® BID (Group A) or matching placebo (Group B) in a 1:1 treatment allocation. Subjects will take the study medications (Theramine® or placebo) for the duration of this phase and complete daily headache diaries. Participants will also complete a Headache Impact Questionnaire (HIT-6), which is a validated questionnaire to assess headache related disability in the last month. This phase will not be included in the data analysis as it may take 1 month to see a treatment effect after starting a preventative.

Phase 3: Phase 3 will last 2 months and represents the time period during which the efficacy of Theramine® will be determined. Participants will continue to complete headache diaries and will continue to Theramine® or placebo during this phase. They will also complete a HIT-6 questionnaire.

There will be four study visits, which will be described below.

Office Visit 1: Following informed consent, a physical and neurological exam and vital signs will be completed. A urine or serum pregnancy test will be collected by all female subjects of childbearing potential. Routine labs (electrolyte panel with creatinine, liver enzyme profile and CRP), will be collected. Eligible participants will be trained during the visit to complete daily headache diaries. It is anticipated that this visit will last for 2 hours.

Office Visit 2: At Visit 2, research staff will review the diary information completed during phase 1. Subjects who complete a minimum of 25 out of 30 days of their daily headache diary will be asked to continue participation with Phase 2 of the study. They will receive 268 capsules of study medication (enough for 67 days) and will be instructed to record any adverse events experienced from taking the study medication. During the office visit, subjects will complete the HIT-6 questionnaire. It is anticipated that this visit will last for 1 hour.

Office Visit 3: At Visit 3, research staff will review the diary information completed during phase 1. Subjects who complete a minimum of 50 out of 60 days of their daily headache diary and took 80% of their study medication will be asked to complete the last month of the study. They will receive 134 capsules of study medication (enough for 33 days) and will be instructed to record any adverse events experienced from taking the study medication. During the office visit, subjects will complete the HIT-6 questionnaire. It is anticipated that this visit will last for 1 hour.

Office Visit 4: At Visit 4, medical and medication history will be updated and adverse events collected. A urine or serum pregnancy test will be collected by any subjects of childbearing potential if study medication was taken and a blood test for CRP will be done. Pregnancy testing and CRP may be completed at Visit 3 if subjects will not be returning for a Visit 4. Study medication accountability and compliance will be assessed by counting all the pills that had been returned by the study participant. Subjects will complete the HIT-6 questionnaire. It is anticipated that this visit will last for 1 hour.

The study coordinator will contact participants by phone, email, mail or texting at least one time per month to schedule appointments and discuss any questions. This study is minimal risk and subjects will not need to return study drug if they withdraw or are withdrawn by the investigator. Information regarding study medication that is not returned for any reason will be documented in the study medication accountability log. Lost to follow up will be defined as any subject who has failed to contact the study coordinator after the coordinator has made six attempts to contact the subject over a 30 day period.

The Investigator will access in a case-by-case basis should a subject request additional days to complete the study or request replacement study medication due to loss. Documentation of such requests and outcomes will be maintained in subject's study file.

ELIGIBILITY:
INCLUSION CRITERIA: The inclusion criteria will be the following:

1. (male and female) 18-65 years of age
2. Women of child-bearing potential, has a negative pregnancy test (urine or serum) at screen, and agrees to one of the following:

   1. Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval (5 days) after completion or premature discontinuation from the study,
   2. History of bilateral tubal ligation,
   3. Hormonal Contraception (oral, patch, etc.) as approved by the Investigator,
   4. Sterilization of male partner; or,
   5. Any intrauterine device (IUD),
   6. Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or spermicide plus a female diaphragm); or,
   7. Any other barrier methods (only if used in combination with any of the above acceptable methods);
3. Diagnosis of migraine headache (ICHD 1.1-1.5) as determined by criteria established by the International Classification of Headache Disorder (ICHD-II).
4. 4-14 days per month with migraine averaged over past 3 months, as self reported by subject.
5. Migraines symptoms must have been present for at least one year prior to enrollment in the study.
6. The onset of migraine symptoms must have occurred before age 50.
7. Is medically stable as determined by the Investigator.
8. If taking any concomitant preventative medication(s), is on a stabilized dosage at the discretion of the investigator.
9. Is willing to stay on current preventative medication(s) for the duration of the study.
10. Is able to take oral medication, adhere to the medication regimens and perform study procedures.
11. Is able to understand and communicate intelligibly with the study observer.
12. Is able to read and comprehend written instructions and be willing to complete all procedures and assessments required by this protocol.
13. Is able to demonstrate the willingness to participate by signing and understanding an informed consent after full explanation of the study.

EXCLUSION CRITERIA: The exclusion criteria will be the following:

1. Is pregnant, actively trying to become pregnant, or breast feeding.
2. A diagnosis of medication overuse headaches as determined by the investigator.
3. Chronic medical illnesses (eg. lupus, malignancy, infections, sarcoidosis) that could potentially modulate the frequency of migraine headache.
4. Has evidence of alcohol or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
5. Chronic daily headache (≥ 15 days per month with headache of any kind) averaged over past 3 months.
6. Abnormal creatinine, BUN, and/or Liver Function Enzymes will be assessed and exclusion will be at the discretion of the Investigator.
7. Allergy or hypersensitivity to any ingredients in Theramine® including arginine-containing preparations and whey protein (milk).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Martin, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Cincinnati Physicians Company, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Blinding information is not available from Funder, but should it become available results will be updated.
Groups:
- All Participants: 2 capsules before breakfast and dinner (BID) for 16 weeks.
  Migraine preventative medications will be permitted, but no changes in dosage will be allowed during the four month study. Migraine abortive meds will be permitted and will be administered per their standard routine.
  Theramine (medical food/old drug): Theramine® is a prescription medical food that is composed of variety of amino acids and/or their precursors.
  Placebo (l-alanine): Theramine like placebo comparator
Period: Overall Study
Arm/Group | All Participants
Started | 31
Completed | 24
Not Completed | 7
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 44.8 [22 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 18
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Migraine/Headache Days
Description: The primary outcome measure will be the frequency of migraine and all headache days in the Theramine active group versus the Theramine placebo group during the treatment period.
Time Frame: 4-6 months
Population: Study funding ended prematurely. Blinding information not provided by Funder. Data analysis was not completed.
Groups:
- Theramine: 2 capsules before breakfast and dinner (BID) for 16 weeks.
  Migraine preventative medications will be permitted, but no changes in dosage will be allowed during the four month study. Migraine abortive meds will be permitted and will be administered per their standard routine.
  Theramine (medical food/old drug): Theramine® is a prescription medical food that is composed of variety of amino acids and/or their precursors.
- Placebo (L-alanine): 2 capsules before breakfast and dinner (BID) for 16 weeks.
  Migraine preventative medications will be permitted, but no changes in dosage will be allowed during the four month study. Migraine abortive meds will be permitted and will be administered per their standard routine.
  Placebo (l-alanine): Theramine like placebo comparator
Arm/Group | Theramine | Placebo (L-alanine)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change in Migraine and Headache Frequency
Description: The percent change in migraine and headache frequency will be defined as [frequency/baseline phase - frequency/treatment phase] divided by [frequency/baseline phase].
Time Frame: 4-6 months
Population: Study funding ended prematurely. Blinding information not provided by Funder. Data analysis was not completed.
Arm/Group | Theramine | Placebo (L-alanine)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: HIT-6
Description: Differences in the scores for the HIT-6 disability inventory between baseline and the last study visit will be analyzed.
Time Frame: 4-6 months
Population: Study funding ended prematurely. Blinding information not provided by Funder. Data analysis was not completed.
Arm/Group | Theramine | Placebo (L-alanine)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Blinding information is not available from Funder. Data analysis was not completed and adverse event terms for non-serious adverse events are only available by Organ System.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=31)
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1) — Not related to study treatment
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=31)
Infections and Infestations (Infections and infestations) | 4 (4)
Nervous System Disorder (Nervous system disorders) | 5 (5)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3)
Gastrointestinal Disorders (Gastrointestinal disorders) | 9 (9)
General Disorders (General disorders) | 1 (1)
Skin and subcutaneious tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3)
Eye Disoders (Eye disorders) | 2 (2)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Metabolism and nutritional disorders (Metabolism and nutrition disorders) | 1 (1)
Reproductive system and breast disoders (Reproductive system and breast disorders) | 1 (1)
Surigical and Medical Procedures (Surgical and medical procedures) | 1 (1) — Elective surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes